CLINICAL TRIAL: NCT07168954
Title: Smart Light Therapy Glasses for Sleep and Mental Wellness, A Randomized Controlled Trial
Brief Title: Smart Light Therapy Glasses for Sleep and Mental Wellness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Waterloo (Other)
Collaborators: Lumos Health Inc. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 43406
Record Dates: First submitted 2025-09-04; First posted 2025-09-11 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-08

CONDITIONS: Depression; Sleep Disturbance
MeSH Terms: conditions — Depression; Parasomnias

STUDY DESIGN:
Intervention Model Description: The intervention group receives full dose light therapy for the full 8 weeks. The control group receives placebo light therapy from week 1 to week 4, followed by full dose light therapy from week 4 to week 8
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Fully blinded study with participants and clinical assessment team blinded. Investigators and outcome assessors access only coded data that masks the interventional after the study to perform analysis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Active Comparator): The treatment group receives fully operational light therapy glasses, with an optimal light output of 500-700 melanopic lux during full power. The users are recommended to wear the glasses for as long as possible during the day, with a minimum requirement of 20 minutes per day. After 8 weeks, this group is cross-overed to receive the placeobo (low dose 50-70 melanopic lux) treatment for another 8 weeks.
  Interventions: Device: Lumos Glasses
- control group (Placebo Comparator): The control group receives placebo operational light therapy glasses, operating at 50-70 melanopic lux during full power. The users are recommended to wear the glasses for as long as possible during the day, with a minimum requirement of 20 minutes per day.
  At week 8, the glasses ramp up to the full 500-700 melanopic lux and becomes equivalent to the active comparator group.
  Interventions: Device: Lumos Glasses

INTERVENTIONS:
Device: Lumos Glasses — The Lumos Glasses provided tailored blue light therapy and blue light filtering based on the time of day and the user's ambient light conditions. It combines the effect of bright blue light therapy and blue light blocking.

SUMMARY:
A pair of smart light therapy glasses (Lumos Glasses) was engineered to control the amount of blue light exposure at a person's eyes through a battery powered light source and nano-coating that reflect blue light.

The research aims to study the effects of this pair of light therapy glasses on depression and sleep.

In addition, the research aims to study the effects of duration of use and its correlation with depression and sleep improvements.

DETAILED DESCRIPTION:
Light has a fundamental impact on human biology. Bright light triggers photoreceptors at the back of the retina to induce neurobiological changes in the brain, affecting neurotransmitter levels such as melatonin and cortisol. For those struggling with depression and sleeping disorders, medical professionals generally recommend the use of a light therapy lamp for 30 minutes a day and the patient begins to improve within the first few weeks of use. However, due to the practical limitations of current light therapy devices such as lamps and head gears, longer durations (2 hours or more) of light therapy each day are often considered infeasible for a modern person, and even adherence to 30 minute are low. As such, the correlation of light therapy duration on sleep and mood improvements are not well understood. Due to this hardware limitation, many research efforts aim to study methods to reduce the duration of light therapy for practical benefits, leading to significant limitations and bias in the understanding of light therapy as well as its clinical implications.

From an alternate perspective of understanding, while the intensity of light from a light therapy box (5000 - 10 000 lux) is brighter than average indoor conditions (500 lux), it rarely exceeds the brightness of light from natural outdoors (up to 100 000 lux). And research also suggests that spending time outdoors could be just as effective as a method as light therapy in treating seasonal affective disorder. As such, it is possible that light therapy's role is to make up for a lack of natural light exposure. In this paper, it is hypothesized that the optimal benefits for light therapy can be achieved by simulating light conditions from natural daylight, on average 12 hours of bright light exposure during the day and 12 hours of no light at night. To validate this theory, a consumer friendly light therapy glasses using an innovative nano coating was engineered to allow for full day unencumbered usage.

The Lumos Glasses' nano-coating design is a state of the art advancement in the light therapy wearable space. LED light sources mounted on the side legs (temples) of the glasses project a band of wavelengths of light centred around 480nm (most impactful for neurobiology based on melanopsin response) onto the nano-coating of the glasses, which is designed to reflect only this specific band of light back into the eyes of the user. This design allows the user to be able to see the world through a regular looking pair of glasses while receiving light therapy. The nano-coating, by design, also filters out 480nm band light from the external environment, thus allowing the glasses to be used as blue light blocking glasses in the evenings when the LEDs are off. Due to the geometry of reflection, the light from the glasses enters at an angle of approximately 35 degrees into the user's eyes. This design is unique in that it is able to miss the fovea region of the eye, allowing for less obstructing of vision, while still activating the ganglion cells which are responsible for photobiology.

Because of the unique light delivery method, it is important that the clinical effect of light therapy through the method of angular light delivery through the nano-coating on glasses is validated. The first objective study is to validate the functional effect of the glasses on depression and sleep improvements through a double blind placebo controlled trial.

In the trial, participants are obligated to wear the glasses for 30 minutes a day, however, are strongly recommended to wear it for longer based on the hypothesis above (up to 12 hours during the day following the natural light dark cycle). It is hypothesized that longer durations of usage (matching the natural cycle) would lead to better results. Thus, the second objective of the study is to observe the distribution of adherence and usage time of the glasses in the study population, as well as determine the correlation between average duration of usage and depression and sleep score improvements.

ELIGIBILITY:
Inclusion:

Adults, any gender, 18+ years old, residing in Ontario Montgomery Asberg Depression Rating Scale Score > 7 or PROMIS score >25 Spend on average less than 2 hours outdoors daily.

Exclusion Criteria:

MADRS Score above 45, or MADRS suicide score is 5 or 6 People with eye disorders or previous eye surgeries. People who have cataracts, macular degeneration, diabetic retinopathy, or other eye disorders. People taking light sensitizing medication. People with bipolar, psychotic disorders or a history of these disorders. People with epilepsy, or history of epilepsy. People with electronic implants, such as pacemakers. Prescription glasses wearers, except for people who can self-supply contact Page 6 of 40 lenses for the duration of the study. People who do not have an iOS or Android based smartphone Shift workers who work night shift or rotating shifts with night shifts

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2024-09-03 (Actual); Primary Completion 2025-07-14 (Actual); Study Completion 2025-07-14 (Actual)

PRIMARY OUTCOMES:
Montgomery Asberg Depression Rating Scale (MADRS) Improvements | 8 weeks, assessed by clinical team at week 0, 4 and 8
  Improvement of depression rating post intervention
PROMIS-Sleep Disturbance-Short Form | 8 weeks, assessed by clinical team at week 0, 4 and 8, self assessed at week 1, 2 ,3, 5, 6, 7
  Improvement of patient reported sleep rating post intervention

SECONDARY OUTCOMES:
Reaction Time Test | 8 weeks, self assessed weekly via the smartphone app at 8pm
  Reaction time test using the smartphone based Psychomotor Vigilance Task
Memory test | 8 weeks, self assessed weekly via the smartphone app at 8pm
  Paired word test using the smartphone

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan M Oakman, Phd, Psychology, Principal Investigator — University of Waterloo
Locations (1):
- University of Waterloo, Waterloo, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
Anonymized participant data will be shared, along with study protocol and statistical analysis methods
Supporting Information: Study Protocol, SAP, CSR
Time Frame: The data will be available upon publication and will be stored for 25 years
Access Criteria: Open access

REFERENCES:
- See also: Website of the Lumos Glasses product — https://www.lumosglasses.com/